CLINICAL TRIAL: NCT01829737
Title: Epidemiologic Studies of Plasmodium Falciparum Gametocytemia and Transmission-blocking Immunity in Kenieroba, Mali
Brief Title: Malaria Transmission Studies in Mali
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Faculty of Science and Technology - FST (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999913107; 13-I-N107
Record Dates: First submitted 2013-04-09; First posted 2013-04-11 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2015-01-20

CONDITIONS: Malaria, Falciparum
Keywords: Asymptomatic Parasitemia; RBC Polymorphism; Acquired Immunity
MeSH Terms: conditions — Malaria, Falciparum

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Malaria is an illness caused by a parasite spread by mosquitoes. When a mosquito bites a person who is infected with a kind of parasite called a gametocyte, it is able to spread the infection to another person. Not everyone infected with parasites have gametocytes in their blood. As a result, not everyone can spread malaria to others. Researchers are interested in learning more about why some healthy people have gametocytes in their blood and others do not. Identifying the people who have gametocytes in their blood can help target treatment and reduce the spread of malaria. This study will focus on the people of the village of Kenieroba in Mali, where malaria is common.

Objectives:

- To study the relationship between gametocytes and malaria transmission in Mali.

Eligibility:

- Individuals between 6 months and 65 years of age who live in Kenieroba, Mali, and will stay in the area for 1 year.

Design:

* For 1 year, participants will have study visits once every 2 weeks (twice a month, for a total of 24 visits). The visits will last 30 minutes each.
* At each visit, participants will provide a small blood sample. They will report any symptoms of malaria such as fever, headache, and body aches. Participants will be encouraged to seek medical treatment if they experience malaria symptoms between visits.
* Participants who have malaria symptoms will have a blood test for malaria parasites. Those who have parasites in the blood will receive antimalarial treatment.
* Three times over 1 year, a larger blood sample will be collected. These blood samples will be taken once in the dry season, once in the wet season, and once in the next dry season.
* Women between 14 and 45 years of age will also provide urine samples to test for pregnancy. Pregnant women will not be asked to give blood samples.

DETAILED DESCRIPTION:
Plasmodium falciparum malaria continues to evade control efforts in part through the complexity of its life cycle, which involves both humans and mosquitoes. While it is known that the gametocyte form of the parasite transmits disease, it is unclear which individuals constitute the primary gametocyte reservoir in a given human population. It is also unclear how an individual s asexual parasite density, acquired immune responses, and red blood cell (RBC) polymorphisms affect the presence and transmission of gametocytes. Investigating these effects has been limited in part because gametocytes are often present in peripheral blood at densities below the limit of microscopic detection. Recent technical advances in the molecular detection of gametocytes have set the stage for a better understanding of gametocyte epidemiology and biology in humans. In a setting of highly seasonal transmission, we are conducting an epidemiological study to estimate gametocyte prevalence over 1 year in the village of Kenieroba, Mali. In a cohort of 500 individuals that represents the age-distribution of the entire village population, we will explore how age, asexual parasite prevalence, season, and RBC polymorphisms affect variation in gametocyte prevalence (detected by a sensitive molecular method). From these same individuals, we will purify plasma IgG and compare its transmission-blocking activity by age group and season. These assessments will provide a foundation for future studies of gametocytemia dynamics within individuals as well as the impact of host immunity on gametocyte infectivity in our study population. Such information will enable us to identify those individuals that are primarily responsible for malaria transmission in Kenieroba. Incorporation of such findings into new or existing computer-based models of parasite infection and transmission may improve our evaluation of existing malaria control strategies.

ELIGIBILITY:
* INCLUSION CRITERIA (COHORT STUDY)

  1. Age 6 months to 65 years, inclusive
  2. Resident of Kenieroba with no plans to relocate away from Kenieroba for 1 year
  3. Willingness to participate in the study as evidenced by informed consent (if <18 years, the informed consent of parent or guardian of the child, and assent from children 14 to 17 years old)

EXCLUSION CRITERIA (COHORT STUDY)

1. Any condition that in the opinion of the investigator would render the participant unable to comply with the protocol (e.g., psychiatric disease)
2. Any health condition that in the opinion of the investigator would confound data analysis or pose unnecessary exposure risks to study personnel (e.g., individuals who are known to be HIV-infected) or to the participant (e.g., severe malnutrition)
3. Pregnancy for venous blood collections (March 2013, October 2013, March 2014)

INCLUSION CRITERIA (ADULT BLOOD COLLECTION STUDY)

1. Age 18 to 65 years, inclusive
2. Hb level greater than or equal to 8.5 g/dL
3. Willingness to participate in the study as evidenced by informed consent

EXCLUSION CRITERIA (ADULT BLOOD COLLECTION STUDY)

1. Pregnancy
2. Any condition that in the opinion of the investigator would render the participant unable to comply with the protocol (e.g., psychiatric disease)
3. Any health condition that in the opinion of the investigator would confound data analysis or pose unnecessary exposure risks to study personnel (e.g., individuals who are known to be HIV-infected) or to the participant (e.g., severe malnutrition)

INCLUSION CRITERIA (PARASITIZED BLOOD COLLECTION STUDY):

1. Age 2 to 17 years, inclusive
2. Hb level greater than or equal to 8.5 g/dL
3. Previous enrollment in cohort study on protocol #08-I-N120
4. Uncomplicated malaria*
5. P. falciparum density greater than or equal to 10,000/microliters
6. Known hemoglobin type HbAA or HbAS
7. Not enrolled in this protocol s cohort study
8. Willingness to participate in the study as evidenced by informed consent and assent from children 14-17 years old)

   * Uncomplicated malaria: axillary temperature >37.5 degrees Celcius or history of fever in the past few days and no criteria of SM (see next paragraph) and no other etiologies of febrile illness (e.g., respiratory tract infection) on clinical examination.

Severe P. falciparum malaria: parasitemia of any density and any one of the following: coma

(Blantyre coma score less than or equal to 2), convulsions (witnessed by investigator), severe prostration, severe anemia (hemoglobin less than or equal to 6 g/dl), respiratory distress, hypoglycemia (serum glucose less than or equal to less than or equal to 40 mg/dl), jaundice/icterus, shock (systolic blood pressure less than or equal to 70 mmHg, rapid pulse, cool extremities), cessation of eating and drinking, repetitive vomiting.

EXCLUSION CRITERIA (PARASITIZED BLOOD COLLECTION STUDY):

1. Pregnancy
2. Any condition that in the opinion of the investigator would render the participant unable to comply with the protocol (e.g., psychiatric disease)
3. Any health condition that in the opinion of the investigator would confound data analysis or pose unnecessary risks to study participants (e.g., severe malnutrition, acquired or inherited immunodeficiency)

Ages: 6 Months to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 534 (Actual)
Dates: Start 2013-03-20; Primary Completion 2015-01-20 (Actual); Study Completion 2015-01-20 (Actual)

PRIMARY OUTCOMES:
Determine gametocytemia prevalence at each time point relative to age group, asexual parasitemia prevalence, season, and red blood cell polymorphisms, for all cohort enrollees residing in Kenieroba and not treated for malaria during the previous... | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Rick M Fairhurst, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Baker DA. Malaria gametocytogenesis. Mol Biochem Parasitol. 2010 Aug;172(2):57-65. doi: 10.1016/j.molbiopara.2010.03.019. Epub 2010 Apr 8. PMID 20381542
- [Background] Sachs J, Malaney P. The economic and social burden of malaria. Nature. 2002 Feb 7;415(6872):680-5. doi: 10.1038/415680a. PMID 11832956
- [Background] Marsh K. Research priorities for malaria elimination. Lancet. 2010 Nov 13;376(9753):1626-7. doi: 10.1016/S0140-6736(10)61499-7. Epub 2010 Oct 28. No abstract available. PMID 21035843
- [Derived] Willcox AC, Huber AS, Diouf A, Barrett JR, Silk SE, Pulido D, King LDW, Alanine DGW, Minassian AM, Diakite M, Draper SJ, Long CA, Miura K. Antibodies from malaria-exposed Malians generally interact additively or synergistically with human vaccine-induced RH5 antibodies. Cell Rep Med. 2021 Jun 21;2(7):100326. doi: 10.1016/j.xcrm.2021.100326. eCollection 2021 Jul 20. PMID 34337556